CLINICAL TRIAL: NCT06493370
Title: Intravenous Ascorbate Plus Gemcitabine/Carboplatin: A Novel and Cost-Effective Alternative With Evident Efficacy in Patients With Muscle Invasive Bladder Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, John Taylor, Director of Basic Urologic Research, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2024-IVC GC MIBC
Record Dates: First submitted 2024-06-26; First posted 2024-07-10 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2024-07

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: This phase 2 study is not randomized or blinded. All eligible participants will be enrolled to avoid bias and be evaluated for adverse events. Due to the small sample size, patients who do not complete neo-adjuvant therapy will be evaluated for toxicity but maybe replaced for efficacy analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intravenous ascorbic acid/vitamin C (Experimental): 2 Cycles Carboplatin Day 1 and Gemcitabine Days 1 and 8 (NAC)
  + Intravenous Vitamin C Days 1-28
  Interventions: Drug: Intravenous ascorbic acid/vitamin C

INTERVENTIONS:
Drug: Intravenous ascorbic acid/vitamin C — A dose escalation regimen will be initiated for each participant at a single dose of 25 g, titrated to up target peak plasma concentration. Once established, IVC will be administered intravenously 2 times per week for the remaining cycles

SUMMARY:
This is a phase II, single arm, Simon two-stage design, trial, enrolling patients with cisplatin ineligible MIBC and/or those patients who decline cisplatin based NAC.

Assess rates of pathologic downstaging and quality of life in MIBC cisplatin-ineligible/declined patients when IVC is added to gemcitabine-carboplatin NAC.

DETAILED DESCRIPTION:
The investigator has hypothesized adding IVC to carbo/gem NAC will enhance pathological downstaging and improve QOL. The patients eligible for this study (cisplatin ineligible or declined with MIBC) typically proceed straight to cystectomy within 12 weeks of initial diagnosis.

In this study, participants will receive two cycles of gemcitabine/carboplatin, along with IVC and then proceed to cystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Ability of participant to understand this study, and participant willingness to sign a written informed consent
* Consent to participate in biorepository protocol number GUB-BCR-001, KU IRB Approved HSC # STUDY00141546
* Males and females age ≥ 18 years
* ECOG Performance Status (PS) 0 - 2
* Women of childbearing potential must have a negative serum pregnancy test 72 hours prior to initiating treatment.
* Diagnosis/disease status Cisplatin-ineligible or declined muscle invasive bladder cancer. Cisplatin ineligibility will be defined based on Galsky criteria: CTCAE ver. 5.0 Grade 2 or greater peripheral neuropathy; CTCAE ver. 5.0 Grade 2 or greater hearing loss; Creatinine clearance estimated or calculated < 60 ml/min; NYHA class II or greater congestive heart failure
* Adequate organ function, defined as follows: Absolute Neutrophil Count >1.5K/UL. (NOTE: Patients with established diagnosis of benign neutropenia are eligible to participate with ANC between 1000-1500 based on discretion of the treating physician.); Platelets >100K/UL; Hemoglobin ≥ 9 g/dL; Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or calculated creatinine clearance ≥ 30 mL/min using the Cockcroft-Gault equation; Total bilirubin ≤ 2.0 x ULN; Aspartate aminotransferase (AST [SGOT]) and alanine aminotransferase (ALT [SGPT]) ≤ 2.5 x ULN unless liver metastases are present, in which case they must be ≤ 5 x ULN; Normal Glucose-6-phosphate dehydrogenase (G6PD) status
* Women of child-bearing potential (WOCBP) and men with partners of child-bearing potential must agree not to donate sperm (men), to practice sexual abstinence or to use the forms of contraception listed in Child-Bearing Potential/Pregnancy section for the duration of study participation and for WOMEN: 6 months after EOT, MEN: 3 months after EOT following completion of therapy.

Exclusion Criteria:

* Simultaneously enrolled in any therapeutic clinical trial
* Current or anticipating use of other anti-neoplastic or investigational agents while participating in this study
* Diagnosed with a psychiatric illness or is in a social situation that would limit compliance with study requirements
* Is pregnant or breastfeeding. There is a potential for congenital abnormalities and for this regimen to harm breast feeding infants
* Women of childbearing age expecting to conceive children while receiving study treatment and for 6 months after the last dose of study treatment. Men expecting to conceive children while receiving study treatment and for 3 months after the last dose of study treatment
* Has a severe known allergic reaction to any excipient contained in the study drug formulation
* Active Grade 3 or 4 (per the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0109) viral, bacterial, or fungal infection within 2 weeks prior to the first dose of study treatment.
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, as determined per treating physician.
* Histology of pure adenocarcinoma, pure squamous cell carcinoma, or pure small cell carcinoma in the TURBT sample
* Current consumption of tobacco products, patients may be asked to quit for 2 weeks prior to enrollment
* If tobacco use is suspected at any point during the trial, cotinine level will be obtained
* History of G6PD deficiency
* History of oxalate renal calculi - per discretion of treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Post treatment pathological staging | Approximately 10 to 12 weeks
  To assess pathologic downstaging rate in MIBC cisplatin-ineligible patients when IVC is added to a gemcitabine/carboplatin NAC regimen. Pre and Post treatment specimen pathology results evaluated per American Joint Committee on Cancer (AJCC) staging guidelines.

SECONDARY OUTCOMES:
To assess Quality of life (QOL) | Approximately 10 to 16 weeks
  Overall change in participant-reported quality of life outcomes. Fact-Bladder (FACT-BI) Quality of life questionnaire as measurement tool.
To measure Disease Free Survival (DFS) | Approximately 2 years
  Disease free survival rate (DFS) among participants
To measure Disease Specific Survival (DSS) | Approximately 2 years
  Disease specific survival rate among participants

OTHER OUTCOMES:
Cellular outcome markers, IVC uptake, IVC specific mechanism markers, Cell death, Cell proliferation | During surgery
  Tumor samples will be collected at timepoints as listed in the protocol study procedures and schedule of events table for evaluation of generally used cellular outcome markers, as well as markers for IVC specific mechanism, via the IRB approved BCa tumor bank (Taylor PI). Acetylated tubulin levels and transferrin receptor levels in tumor samples will be detected as IVC related markers. SLC23A2 (SVCT2, vitamin C tissue receptor) will be assessed for drug uptake. TUNEL staining will be used as a measure of cell death and Ki67 as a measure of cell proliferation. Circulating tumor DNA (ctDNA) will be assessed in serum as an additional marker of treatment efficacy and recurrence. In addition, single-cell sequencing will be used to define changes in specific tissue populations at TUR and RC to evaluate both biomarkers of response and potential mechanisms associated with IVC treatment. To monitor inflammation, urinary cytokines will be assessed via multiplex ELISA at RC (post-treatment).

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Holden Comprehensive Cancer Center - The University of Iowa, Iowa City, Iowa
  - The University of Kansas Cancer Center, Kansas City, Kansas

REFERENCES:
- [Background] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835
- [Background] Kamat AM, Hahn NM, Efstathiou JA, Lerner SP, Malmstrom PU, Choi W, Guo CC, Lotan Y, Kassouf W. Bladder cancer. Lancet. 2016 Dec 3;388(10061):2796-2810. doi: 10.1016/S0140-6736(16)30512-8. Epub 2016 Jun 23. PMID 27345655
- [Background] Hermans TJN, Voskuilen CS, van der Heijden MS, Schmitz-Drager BJ, Kassouf W, Seiler R, Kamat AM, Grivas P, Kiltie AE, Black PC, van Rhijn BWG. Neoadjuvant treatment for muscle-invasive bladder cancer: The past, the present, and the future. Urol Oncol. 2018 Sep;36(9):413-422. doi: 10.1016/j.urolonc.2017.10.014. Epub 2017 Nov 8. PMID 29128420
- [Background] Carles J, Nogue M, Domenech M, Perez C, Saigi E, Villadiego K, Guasch I, Ibeas R. Carboplatin-gemcitabine treatment of patients with transitional cell carcinoma of the bladder and impaired renal function. Oncology. 2000 Jun;59(1):24-7. doi: 10.1159/000012132. PMID 10895062
- [Background] Sternberg CN, Bellmunt J, Sonpavde G, Siefker-Radtke AO, Stadler WM, Bajorin DF, Dreicer R, George DJ, Milowsky MI, Theodorescu D, Vaughn DJ, Galsky MD, Soloway MS, Quinn DI; International Consultation on Urologic Disease-European Association of Urology Consultation on Bladder Cancer 2012. ICUD-EAU International Consultation on Bladder Cancer 2012: Chemotherapy for urothelial carcinoma-neoadjuvant and adjuvant settings. Eur Urol. 2013 Jan;63(1):58-66. doi: 10.1016/j.eururo.2012.08.010. Epub 2012 Aug 14. PMID 22917984
- [Background] Ma Y, Chapman J, Levine M, Polireddy K, Drisko J, Chen Q. High-dose parenteral ascorbate enhanced chemosensitivity of ovarian cancer and reduced toxicity of chemotherapy. Sci Transl Med. 2014 Feb 5;6(222):222ra18. doi: 10.1126/scitranslmed.3007154. PMID 24500406
- [Background] Polireddy K, Dong R, Reed G, Yu J, Chen P, Williamson S, Violet PC, Pessetto Z, Godwin AK, Fan F, Levine M, Drisko JA, Chen Q. High Dose Parenteral Ascorbate Inhibited Pancreatic Cancer Growth and Metastasis: Mechanisms and a Phase I/IIa study. Sci Rep. 2017 Dec 7;7(1):17188. doi: 10.1038/s41598-017-17568-8. PMID 29215048
- [Background] Espey MG, Chen P, Chalmers B, Drisko J, Sun AY, Levine M, Chen Q. Pharmacologic ascorbate synergizes with gemcitabine in preclinical models of pancreatic cancer. Free Radic Biol Med. 2011 Jun 1;50(11):1610-9. doi: 10.1016/j.freeradbiomed.2011.03.007. Epub 2011 Mar 12. PMID 21402145
- [Background] Du J, Martin SM, Levine M, Wagner BA, Buettner GR, Wang SH, Taghiyev AF, Du C, Knudson CM, Cullen JJ. Mechanisms of ascorbate-induced cytotoxicity in pancreatic cancer. Clin Cancer Res. 2010 Jan 15;16(2):509-20. doi: 10.1158/1078-0432.CCR-09-1713. Epub 2010 Jan 12. PMID 20068072
- [Background] Yun J, Mullarky E, Lu C, Bosch KN, Kavalier A, Rivera K, Roper J, Chio II, Giannopoulou EG, Rago C, Muley A, Asara JM, Paik J, Elemento O, Chen Z, Pappin DJ, Dow LE, Papadopoulos N, Gross SS, Cantley LC. Vitamin C selectively kills KRAS and BRAF mutant colorectal cancer cells by targeting GAPDH. Science. 2015 Dec 11;350(6266):1391-6. doi: 10.1126/science.aaa5004. Epub 2015 Nov 5. PMID 26541605
- [Background] Pollard HB, Levine MA, Eidelman O, Pollard M. Pharmacological ascorbic acid suppresses syngeneic tumor growth and metastases in hormone-refractory prostate cancer. In Vivo. 2010 May-Jun;24(3):249-55. PMID 20554995
- [Background] Monti DA, Mitchell E, Bazzan AJ, Littman S, Zabrecky G, Yeo CJ, Pillai MV, Newberg AB, Deshmukh S, Levine M. Phase I evaluation of intravenous ascorbic acid in combination with gemcitabine and erlotinib in patients with metastatic pancreatic cancer. PLoS One. 2012;7(1):e29794. doi: 10.1371/journal.pone.0029794. Epub 2012 Jan 17. PMID 22272248
- [Background] Welsh JL, Wagner BA, van't Erve TJ, Zehr PS, Berg DJ, Halfdanarson TR, Yee NS, Bodeker KL, Du J, Roberts LJ 2nd, Drisko J, Levine M, Buettner GR, Cullen JJ. Pharmacological ascorbate with gemcitabine for the control of metastatic and node-positive pancreatic cancer (PACMAN): results from a phase I clinical trial. Cancer Chemother Pharmacol. 2013 Mar;71(3):765-75. doi: 10.1007/s00280-013-2070-8. Epub 2013 Feb 5. PMID 23381814
- [Background] Gilloteaux J, Jamison JM, Neal DR, Loukas M, Doberzstyn T, Summers JL. Cell damage and death by autoschizis in human bladder (RT4) carcinoma cells resulting from treatment with ascorbate and menadione. Ultrastruct Pathol. 2010 May;34(3):140-60. doi: 10.3109/01913121003662304. PMID 20455663
- [Background] Chen Q, Espey MG, Krishna MC, Mitchell JB, Corpe CP, Buettner GR, Shacter E, Levine M. Pharmacologic ascorbic acid concentrations selectively kill cancer cells: action as a pro-drug to deliver hydrogen peroxide to tissues. Proc Natl Acad Sci U S A. 2005 Sep 20;102(38):13604-9. doi: 10.1073/pnas.0506390102. Epub 2005 Sep 12. PMID 16157892
- [Background] Chen Q, Espey MG, Sun AY, Lee JH, Krishna MC, Shacter E, Choyke PL, Pooput C, Kirk KL, Buettner GR, Levine M. Ascorbate in pharmacologic concentrations selectively generates ascorbate radical and hydrogen peroxide in extracellular fluid in vivo. Proc Natl Acad Sci U S A. 2007 May 22;104(21):8749-54. doi: 10.1073/pnas.0702854104. Epub 2007 May 14. PMID 17502596
- [Background] Chen Q, Espey MG, Sun AY, Pooput C, Kirk KL, Krishna MC, Khosh DB, Drisko J, Levine M. Pharmacologic doses of ascorbate act as a prooxidant and decrease growth of aggressive tumor xenografts in mice. Proc Natl Acad Sci U S A. 2008 Aug 12;105(32):11105-9. doi: 10.1073/pnas.0804226105. Epub 2008 Aug 4. PMID 18678913
- [Background] Schoenfeld JD, Sibenaller ZA, Mapuskar KA, Wagner BA, Cramer-Morales KL, Furqan M, Sandhu S, Carlisle TL, Smith MC, Abu Hejleh T, Berg DJ, Zhang J, Keech J, Parekh KR, Bhatia S, Monga V, Bodeker KL, Ahmann L, Vollstedt S, Brown H, Kauffman EPS, Schall ME, Hohl RJ, Clamon GH, Greenlee JD, Howard MA, Schultz MK, Smith BJ, Riley DP, Domann FE, Cullen JJ, Buettner GR, Buatti JM, Spitz DR, Allen BG. O2⋅- and H2O2-Mediated Disruption of Fe Metabolism Causes the Differential Susceptibility of NSCLC and GBM Cancer Cells to Pharmacological Ascorbate. Cancer Cell. 2017 Aug 14;32(2):268. doi: 10.1016/j.ccell.2017.07.008. No abstract available. PMID 28810149
- [Background] Deubzer B, Mayer F, Kuci Z, Niewisch M, Merkel G, Handgretinger R, Bruchelt G. H(2)O(2)-mediated cytotoxicity of pharmacologic ascorbate concentrations to neuroblastoma cells: potential role of lactate and ferritin. Cell Physiol Biochem. 2010;25(6):767-74. doi: 10.1159/000315098. Epub 2010 May 18. PMID 20511723
- [Background] Miller DM, Buettner GR, Aust SD. Transition metals as catalysts of "autoxidation" reactions. Free Radic Biol Med. 1990;8(1):95-108. doi: 10.1016/0891-5849(90)90148-c. PMID 2182396
- [Background] Levine M, Conry-Cantilena C, Wang Y, Welch RW, Washko PW, Dhariwal KR, Park JB, Lazarev A, Graumlich JF, King J, Cantilena LR. Vitamin C pharmacokinetics in healthy volunteers: evidence for a recommended dietary allowance. Proc Natl Acad Sci U S A. 1996 Apr 16;93(8):3704-9. doi: 10.1073/pnas.93.8.3704. PMID 8623000
- [Background] Levine M, Wang Y, Padayatty SJ, Morrow J. A new recommended dietary allowance of vitamin C for healthy young women. Proc Natl Acad Sci U S A. 2001 Aug 14;98(17):9842-6. doi: 10.1073/pnas.171318198. PMID 11504949
- [Background] Chen P, Reed G, Jiang J, Wang Y, Sunega J, Dong R, Ma Y, Esparham A, Ferrell R, Levine M, Drisko J, Chen Q. Pharmacokinetic Evaluation of Intravenous Vitamin C: A Classic Pharmacokinetic Study. Clin Pharmacokinet. 2022 Sep;61(9):1237-1249. doi: 10.1007/s40262-022-01142-1. Epub 2022 Jun 25. PMID 35750958
- [Background] Lv H, Wang C, Fang T, Li T, Lv G, Han Q, Yang W, Wang H. Vitamin C preferentially kills cancer stem cells in hepatocellular carcinoma via SVCT-2. NPJ Precis Oncol. 2018 Jan 8;2(1):1. doi: 10.1038/s41698-017-0044-8. eCollection 2018. PMID 29872720
- [Background] Carroll RS, Du J, O'Leary BR, Steers G, Goswami PC, Buettner GR, Cullen JJ. Pharmacological ascorbate induces sustained mitochondrial dysfunction. Free Radic Biol Med. 2023 Aug 1;204:108-117. doi: 10.1016/j.freeradbiomed.2023.04.023. Epub 2023 May 1. PMID 37137343
- [Background] Alexander MS, Wilkes JG, Schroeder SR, Buettner GR, Wagner BA, Du J, Gibson-Corley K, O'Leary BR, Spitz DR, Buatti JM, Berg DJ, Bodeker KL, Vollstedt S, Brown HA, Allen BG, Cullen JJ. Pharmacologic Ascorbate Reduces Radiation-Induced Normal Tissue Toxicity and Enhances Tumor Radiosensitization in Pancreatic Cancer. Cancer Res. 2018 Dec 15;78(24):6838-6851. doi: 10.1158/0008-5472.CAN-18-1680. Epub 2018 Sep 25. PMID 30254147
- [Background] Furqan M, Abu-Hejleh T, Stephens LM, Hartwig SM, Mott SL, Pulliam CF, Petronek M, Henrich JB, Fath MA, Houtman JC, Varga SM, Bodeker KL, Bossler AD, Bellizzi AM, Zhang J, Monga V, Mani H, Ivanovic M, Smith BJ, Byrne MM, Zeitler W, Wagner BA, Buettner GR, Cullen JJ, Buatti JM, Spitz DR, Allen BG. Pharmacological ascorbate improves the response to platinum-based chemotherapy in advanced stage non-small cell lung cancer. Redox Biol. 2022 Jul;53:102318. doi: 10.1016/j.redox.2022.102318. Epub 2022 Apr 20. PMID 35525024
- [Background] Narain TA, Tosh JM, Gautam G, Talwar HS, Panwar VK, Mittal A, Mandal AK. Neoadjuvant Therapy for Cisplatin Ineligible Muscle Invasive Bladder Cancer Patients: A Review of Available Evidence. Urology. 2021 Aug;154:8-15. doi: 10.1016/j.urology.2021.03.010. Epub 2021 Mar 26. PMID 33775784
- [Background] Jain RK, Sonpavde G. Neoadjuvant therapy for muscle-invasive bladder cancer. Expert Rev Anticancer Ther. 2020 Jul;20(7):603-614. doi: 10.1080/14737140.2020.1784011. Epub 2020 Jun 30. PMID 32546025
- [Background] Sadeghi S, Groshen SG, Tsao-Wei DD, Parikh R, Mortazavi A, Dorff TB, Kefauver C, Hoimes C, Doyle L, Quinn DI, Newman E, Lara PN Jr. Phase II California Cancer Consortium Trial of Gemcitabine-Eribulin Combination in Cisplatin-Ineligible Patients With Metastatic Urothelial Carcinoma: Final Report (NCI-9653). J Clin Oncol. 2019 Oct 10;37(29):2682-2688. doi: 10.1200/JCO.19.00861. Epub 2019 Aug 7. PMID 31390274
- [Background] Dogliotti L, Carteni G, Siena S, Bertetto O, Martoni A, Bono A, Amadori D, Onat H, Marini L. Gemcitabine plus cisplatin versus gemcitabine plus carboplatin as first-line chemotherapy in advanced transitional cell carcinoma of the urothelium: results of a randomized phase 2 trial. Eur Urol. 2007 Jul;52(1):134-41. doi: 10.1016/j.eururo.2006.12.029. Epub 2006 Dec 26. PMID 17207911
- [Background] Bellmunt J, Ribas A, Eres N, Albanell J, Almanza C, Bermejo B, Sole LA, Baselga J. Carboplatin-based versus cisplatin-based chemotherapy in the treatment of surgically incurable advanced bladder carcinoma. Cancer. 1997 Nov 15;80(10):1966-72. doi: 10.1002/(sici)1097-0142(19971115)80:103.0.co;2-w. PMID 9366300
- [Background] Petrioli R, Frediani B, Manganelli A, Barbanti G, De Capua B, De Lauretis A, Salvestrini F, Mondillo S, Francini G. Comparison between a cisplatin-containing regimen and a carboplatin-containing regimen for recurrent or metastatic bladder cancer patients. A randomized phase II study. Cancer. 1996 Jan 15;77(2):344-51. doi: 10.1002/(SICI)1097-0142(19960115)77:23.0.CO;2-1. PMID 8625244
- [Background] Einerhand SMH, van Dijk N, van Dorp J, de Feijter JM, van Montfoort ML, van de Kamp MW, Schaake EE, Boellaard TN, Hendricksen K, van der Heijden MS, van Rhijn BWG. Survival after neoadjuvant/induction combination immunotherapy vs combination platinum-based chemotherapy for locally advanced (Stage III) urothelial cancer. Int J Cancer. 2022 Dec 1;151(11):2004-2011. doi: 10.1002/ijc.34125. Epub 2022 Jun 10. PMID 35603905
- [Background] Padayatty SJ, Sun H, Wang Y, Riordan HD, Hewitt SM, Katz A, Wesley RA, Levine M. Vitamin C pharmacokinetics: implications for oral and intravenous use. Ann Intern Med. 2004 Apr 6;140(7):533-7. doi: 10.7326/0003-4819-140-7-200404060-00010. PMID 15068981
- [Background] Padayatty SJ, Sun AY, Chen Q, Espey MG, Drisko J, Levine M. Vitamin C: intravenous use by complementary and alternative medicine practitioners and adverse effects. PLoS One. 2010 Jul 7;5(7):e11414. doi: 10.1371/journal.pone.0011414. PMID 20628650
- See also: National Institute of Health/National Cancer Institute - Cancer Therapy Evaluation Program (CTEP). Common Terminology Criteria for Adverse Events (CTCAE). — https://ctep.cancer.gov/protocoldevelopment/electronic_applications/ctc.htm#ctc_60